CLINICAL TRIAL: NCT01755026
Title: Serum and Tissue Cefazolin Concentrations in Patients Undergoing Cesarean Delivery Receiving Two Differing Doses of Pre-operative Cefazolin.
Brief Title: Serum and Tissue Cefazolin Concentrations in Patients Undergoing Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Stitely (Other)
Responsible Party: Sponsor-Investigator, Michael Stitely, Adjunct Associate Professor, West Virginia University
Organization: West Virginia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-22512
Record Dates: First submitted 2011-06-29; First posted 2012-12-21 (Estimated); Results first posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-06

CONDITIONS: Cesarean Delivery; Wound Infection; Obesity
Keywords: Cesarean Delivery; Wound infection; Obesity; Prophylactic antibiotics
MeSH Terms: conditions — Wound Infection; Obesity | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 gram dose of cefazolin (Active Comparator): 2 gram dose of pre-operative cefazolin
  Interventions: Drug: cefazolin
- 4 gram Dose (Experimental): 4 gram dose of pre-operative prophylaxis
  Interventions: Drug: cefazolin

INTERVENTIONS:
Drug: cefazolin — 2 gram dose for pre-operative prophylaxis
  Other Names: Ancef
  Arms: 2 gram dose of cefazolin
Drug: cefazolin — 4 gram dose for pre-operative prophylaxis
  Other Names: Ancef
  Arms: 4 gram Dose

SUMMARY:
Patients undergoing Cesarean delivery (C-Section) with a body mass index of 35 or greater (this BMI number is in the obese range) will be given either 2 grams or 4 grams of an antibiotic before surgery. The antibiotic is intended to prevent infection from the surgery.It is unknown what the best dose for large women is for the usual medicine used for this purpose (an antibiotic medicine called cefazolin).Samples of the tissue just under the skin will be biopsied at the time the incision is made and at the time the cut is stitched or stapled closed. A sample of the muscle of the womb will be taken as the womb is stitched closed after the delivery. Blood tests will be done at the start and end of surgery to test the antibiotic level. A blood sample will be taken from the umbilical cord after the baby has been delivered and the umbilical cord has been cut. The umbilical cord blood sample will be tested for the antibiotic level.These tests will be used to find out if the usual dose of medicine is enough or if more medicine is needed to prevent infection in large women undergoing c-sections.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above
2. Body mass index (BMI) of 35 or greater at the time of the first obstetric clinic visit
3. Undergoing cesarean delivery

Exclusion Criteria:

1. BMI less than 35.
2. Not undergoing Cesarean delivery.
3. Age less than 18 years.
4. Pre-existing infection.
5. Allergy to cephalosporin medications or a history of an anaphylactic reaction to penicillin.
6. Cesarean delivery being performed under emergent circumstances.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H Holls, MD, Principal Investigator — West Virginia University; Michael L Stitely, MD, Study Chair — West Virginia University
Locations (1):
- West Virginia University Hospital, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4 Gram Dose | 2 Gram Dose of Cefazolin
Started | 11 | 12
Completed | 9 | 11
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 Gram Dose | 2 Gram Dose of Cefazolin | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.33 (4.64) | 31.09 (6.46) | 31 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Cefazolin Levels
Description: Cefazolin levels
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: mcg/mL
Arm/Group | 2 Gram Dose of Cefazolin | 4 Gram Dose
Number analyzed (Participants) | 9 | 11
mcg/mL
  Subcutaneous tissue-opening | 18.36 (6.68) | 40.11 (24.1)
  Subcutaneous tissue-closing | 21.73 (16.02) | 34.89 (17.42)
  Plasma concentration at incision | 155.45 (50.97) | 346.16 (166.01)
  Plasma concentration at closure | 83.49 (34.97) | 150.12 (55.54)
  Myometrial levels | 67.18 (13.89) | 146.22 (60.99)
  Umbilical cord blood concentrations | 25.01 (12.03) | 82.23 (43.03)
Statistical Analysis 1: Comparison: 2 Gram Dose of Cefazolin vs 4 Gram Dose; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Net) = 191, Standard Error of Mean 166.01

ADVERSE EVENTS:
Arm/Group | 4 Gram Dose | 2 Gram Dose of Cefazolin
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 1/11 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 Gram Dose (N=11) | 2 Gram Dose of Cefazolin (N=12)
Allergy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Minor skin reaction with starting cefazolin infusion. Administartion of cefazolin stopped with no further concerns and rash on arm resolved without further treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes